CLINICAL TRIAL: NCT02390128
Title: Giving Children the Best Start in Life: the Mothers and Babies at Yorkhill Thyroid Health
Brief Title: Mothers and Babies at Yorkhill Thyroid Health Cohort
Acronym: MABY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Emilie Combet, Lecturer, University of Glasgow
Other Study IDs: 153466
Record Dates: First submitted 2014-11-30; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Function
Keywords: iodine; thyroid; TSH; pregnancy; nutrition; diet
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, blood, hair, breastmilk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mothers and babies: pregnant mothers (UK resident) and their babies (observational, not an intervention)
  Interventions: Other: observational only

INTERVENTIONS:
Other: observational only

SUMMARY:
This is an observational study in pregnant mothers and their newborn babies. The rationale of the study is to examine early markers of the effects of iodine insufficiency during pregnancy on thyroid stimulating hormone (TSH) and thyroglobulin in mother and baby.

DETAILED DESCRIPTION:
Iodine is a critical component of thyroid hormones, which are essential for normal growth, and brain development, most of the latter occurring during fetal life and in the first three years of life. Maternal dietary iodine is the sole source for fetuses and for exclusively breastfed infants. Recent evidence indicates that the UK female population is not iodine sufficient. Thus a significant proportion of UK pregnant women will also be insufficient in dietary iodine with potential harmful consequences for their babies. We wish to investigate the relationship between maternal iodine status (sufficient versus insufficient) in pregnancy, the mode of neonatal feeding (exclusively breast fed vs exclusively formula fed); and the effect this has on the functioning of the newborn baby's thyroid gland, with provision for later cognitive followup assessment. In order to do this, we will determine:

i) the iodine status of the mother during pregnancy and in the immediate postnatal period (dietary and urinary) and the newborn infant (urinary), ii) the thyroid function of the mother (thyroid stimulating hormone, thyroglobulin, T4 in serum during pregnancy, and thyroid stimulating hormone and thyroglobulin in dried blood spots postpartum) and infant (thyroid stimulating hormone in dried blood spots collected during a routine procedure).

Our hypothesis is that babies whose mothers are iodine insufficient will show higher levels of TSH and thyroglobulin than the babies of iodine sufficient mothers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Able to read, write and speak in English
* Attending a Greater Glasgow and Clyde maternity unit

Exclusion Criteria:

* Abnormal pregnancies.
* Mothers with known thyroid disorders.
* Preterm infants (born before 37 completed weeks).
* Multiple births.
* Infants with postnatal problems such as infection or malformation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their newborn baby
Sampling Method: Non-Probability Sample
Enrollment: 697 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
thyroid function of mothers (measurement of TSH and Tg) | up to 38 week gestation
  measurement of TSH and Tg
thyroid function of infant (routine TSH measurement) | Day 4 of life
  routine TSH measurement

SECONDARY OUTCOMES:
Iodine status of mothers (iodine intake and excretion) | up to 38 week gestation
  iodine status defined by iodine intake and excretion
Iodine status of infant (iodine intake and excretion) | Day 4 of life
  iodine status defined by iodine intake and excretion
Iodine level in hair and breastmilk | after birth
  measurement of iodine in hair and breastmilk

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Cizmecioglu, Principal Investigator — University of Glasgow; Emilie Combet, Study Director — University of Glasgow; Jeremy Jones, Principal Investigator — University of Glasgow; Malcolm Donaldson, Principal Investigator — University of Glasgow
Locations (1):
- NHS GGC Community midwifery units, Glasgow, United Kingdom